CLINICAL TRIAL: NCT04062981
Title: Phase 1, Open-Label Study of Carisbamate in Adult and Pediatric Subjects With Lennox-Gastaut Syndrome
Brief Title: Carisbamate Safety Study in Adult and Pediatric Subjects With Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YKP509C002
Record Dates: First submitted 2019-05-30; First posted 2019-08-20 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Lennox Gastaut Syndrome
MeSH Terms: conditions — Lennox Gastaut Syndrome | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Intervention Model Description: Open-Label (OL), multi-center study of carisbamate in subjects with LGS, with safety assessments from Baseline (Visit 1) through early termination (ET)/end of study (EOS) visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort I (Experimental): Subjects ≥ 18 years of age
  These subjects will reach maximum stable dose and continue onto YKP509C002.
  Interventions: Drug: Carisbamate
- Cohort II (Experimental): Subjects 12 to <18 years of age
  These subjects will reach maximum stable dose and continue onto YKP509C002.
  Interventions: Drug: Carisbamate
- Cohort III (Experimental): Subjects 6 to <12 years of age
  These subjects will reach maximum stable dose and continue onto YKP509C002.
  Interventions: Drug: Carisbamate
- Cohort IV (Experimental): Subjects 2 to <6 years of age
  These subjects will reach maximum stable dose and continue onto YKP509C002.
  Interventions: Drug: Carisbamate

INTERVENTIONS:
Drug: Carisbamate — An oral liquid formulation (20 mg/mL) of carisbamate (S-carisbamate)
  Other Names: YKP509

SUMMARY:
Open-label extension study from YKP509C001 to evaluate the safety and tolerability of carisbamate in subjects with Lennox-Gastaut Syndrome (LGS).

DETAILED DESCRIPTION:
Subjects who successfully completed the YKP509C001 study and could benefit from continued exposure to carisbamate.

This is an open-label (OL), multi-center study of carisbamate in subjects with LGS, with safety assessments from Baseline (Visit 1) through the early termination (ET)/end of study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed the YKP509C001 study
* Investigator believes subject could benefit from continued exposure to study drug
* Subjects must continue to meet all of the inclusion criteria from the YKP509C001 study

Exclusion Criteria:

* Subjects must continue to not meet any of the exclusion criteria from the YKP509C001 study
* There are no additional exclusion criteria in this study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Concomitant medication | Up to 20 months
  Safety
12-lead electrocardiograms (ECGs) | Up to 20 months
  Safety
Physical examinations | Up to 20 months
  Safety
Seizure Frequency | Up to 20 months
  An assessment of seizure frequency will be made using a subject/caregiver seizure diary with seizure type and number of daily seizures recorded since the prior visit.

SECONDARY OUTCOMES:
Safety- adverse events | The duration of this OL study will be until carisbamate bas been approved for treatment of LGS and is available by prescription, or development of carisbamate for LGS has stopped, whichever is first. This could occur up to 36 months.
  Adverse events assessment for seriousness (yes, no) severity (mild, moderate, severe), affect on carisbamate dosing (increase,reduced, interrupted, withdrawn, no change) and outcome (recovered/resolved, recovered/resolved with sequelae, recovering/resolving, not recovered/not resolved, fatal or unknown

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, MD, Study Director — SK Life Science, Inc.
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Oregon Health and Science University, Portland, Oregon
  - The University of Utah School of Medicine - Primary Children's Hospital (Primary Children's Medical Center), Salt Lake City, Utah
  - UW Valley Medical Center, Renton, Washington